CLINICAL TRIAL: NCT05320042
Title: 1-Week Dispensing Evaluation of Kalifilcon A Daily Disposable Toric Contact Lenses Compared to Ultra for Astigmatism Contact Lenses
Brief Title: 1-Week Dispensing Evaluation of Kalifilcon A Toric Contact Lenses Compared to Ultra for Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROC2-21-013
Record Dates: First submitted 2022-04-01; First posted 2022-04-11 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- kalifilcon A Daily Disposable Toric (Experimental): kalifilcon A Daily Disposable Toric
  Interventions: Device: kalifilcon A Daily Disposable Toric
- Ultra for Astigmatism Contact Lenses (Active Comparator): Ultra for Astigmatism Contact Lenses
  Interventions: Device: Ultra for Astigmatism Contact Lenses

INTERVENTIONS:
Device: kalifilcon A Daily Disposable Toric — kalifilcon A Daily Disposable Toric
  Arms: kalifilcon A Daily Disposable Toric
Device: Ultra for Astigmatism Contact Lenses — Ultra for Astigmatism Contact Lenses
  Arms: Ultra for Astigmatism Contact Lenses

SUMMARY:
Experienced soft contact lens wearing subjects will be enrolled in this 1-week, confirmatory, randomized, bilateral, 2-way crossover, double masked (subject and investigator), repeated measures, dispensing study. All subjects will be seen for a Screening/Baseline Visit at which informed consent will be obtained and eligibility will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have the capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study.
2. Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | One week
  Mean Binocular logMAR Visual Acuity

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch site 1, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No